CLINICAL TRIAL: NCT04469361
Title: The Effect of Ballet Training on Plantar Venous Pump Activity in Ballerinas
Brief Title: The Effect of Training on Hemodynamic Factors in Ballet Dancer
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2017.129
Record Dates: First submitted 2020-07-02; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2017-02

CONDITIONS: Venous Insufficiency; Foot Drop (Acquired)
MeSH Terms: conditions — Venous Insufficiency; Peroneal Neuropathies | interventions — Supine Position; Standing Position

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ballerinas: Balerina students who have trained at least for 4 years
  Interventions: Other: Navicular drop measurement; Other: Measurement of venous return parameters in supine; Other: Measurement of venous return parameters in standing; Other: measurement of midfoot pressure distrubition
- Female students: Female students with sedentary lifestyle
  Interventions: Other: Navicular drop measurement; Other: Measurement of venous return parameters in supine; Other: Measurement of venous return parameters in standing; Other: measurement of midfoot pressure distrubition

INTERVENTIONS:
Other: Navicular drop measurement — The difference in navicular height between sitting and standing positions was recorded (mm) as the amount of navicular drop.
Other: Measurement of venous return parameters in supine — Venous return parameters of posterior tibial vein was measured when participant applied force equivalent to their own body weight on plantar surface of their right leg in supine position
Other: Measurement of venous return parameters in standing — In standing, venous return parameters was measured of posterior tibial vein when participants shift all of their weight to the right leg for 3 second with their leg muscles as relaxed as possible and their knee joint in full extension.
Other: measurement of midfoot pressure distrubition — In standing, midfoot pressure distrubution was measured when participants shift all of their weight to the right leg

SUMMARY:
Classic ballet dance is a demonstration of complex motor skills to be revealed in aesthetic combinations and repetitively, and it demands intensive use of the lower extremities within extreme of range of motion (ROM). Because ballet practice depends on advanced technical skills, it involves intensive physical training and causes an overload on the musculoskeletal system and foot deformities such as pes planus.

Plantar venous pump (PVP) is a network of multiple venous vessels located between the muscles of the foot arch. PVP is considered the first step of venous return and discharges into the posterior tibial vein (PTV). PVP is reported to be active during gait while it is inactive in resting position. There are different views on the mechanisms enabling its activation 1-3. The general view is that during the stance phase of the gait, the flattening of the plantar arch with weight transfer causes the veins in this region to narrow and creates a force that pumps the blood up.

The aim of this study is the investigation what kind of hemodynamic changes ballet training causes in the lower extremity

ELIGIBILITY:
Inclusion Criteria (for balerinas):

* receiving ballet training at least 10 h per week for at least 4 years
* receiving formal dancing training system

Inclusion Criteria (for non-dancer group)

* never receiving formal dancing training
* having sedentary lifestyle

Exclusion Criteria:

* Participants with a history of foot or ankle surgery,
* Participants with connective tissue disease,
* Participants with rigid pes planus-cavus,
* Participants with chronic venous insufficiency
* Participants with acute ankle injury in recent 3 months

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — ballerinas and females students with sedentary life styles
Study Population: Ballerinas taking ballet training at least for 4 years and female sedentary students
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of navicular drop | Cchange from baseline navicular height in pre-intervention and immediately after the intervention/
  Navicular drop was measured in mm
Evaluation of diameter of tibialis posterior vein in supine | Change from baseline diameter of tibialis posterior vein during intervention
  Diameter of tibialis posterior vein was measured in mm
Evaluation of flow velocity of tibialis posterior vein in supine | Change from baseline flow velocity of tibialis posterior vein during intervention
  Flow velocity of tibialis posterior vein was measured in cm/s
Evaluation of volume flow of tibialis posterior vein in supine | Change from baseline volume flow of tibialis posterior vein during intervention
  Volume flow of tibialis posterior vein was measured in ml/min
Evaluation of diameter of tibialis posterior vein during weight bearing | Change from baseline diameter of tibialis posterior during intervention
  Diameter of tibialis posterior vein was measured in mm
Evaluation of flow velocity of tibialis posterior vein during weight bearing | Change from baseline flow velocity of tibialis posterior vein during intervention
  Flow velocity of tibialis posterior vein was measured in cm/s
Evaluation of volume flow of tibialis posterior vein during weight bearing | Change from baseline volume flow of tibialis posterior vein during intervention
  Volume flow of tibialis posterior vein was measured in ml/min
Evaluation of midfoot plantar pressure during weight bearing | Change from baseline midfoot pressure during intervention
  Midfoot plantar pressure was measured in gr/cm2

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Kablan, PhD, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guss-West C, Wulf G. Attentional Focus in Classical Ballet: A Survey Of Professional Dancers. J Dance Med Sci. 2016 Mar;20(1):23-9. doi: 10.12678/1089-313X.20.1.23. PMID 27025449
- [Result] Allen N, Nevill A, Brooks J, Koutedakis Y, Wyon M. Ballet injuries: injury incidence and severity over 1 year. J Orthop Sports Phys Ther. 2012 Sep;42(9):781-90. doi: 10.2519/jospt.2012.3893. Epub 2012 Jul 19. PMID 22814244
- [Result] Gardner AM, Fox RH. The venous pump of the human foot--preliminary report. Bristol Med Chir J. 1983 Jul;98(367):109-12. No abstract available. PMID 6616290
- [Result] Kim TI, Forbang NI, Criqui MH, Allison MA. Association of foot and ankle characteristics with progression of venous disease. Vasc Med. 2015 Apr;20(2):105-11. doi: 10.1177/1358863X14568443. PMID 25832598
- [Result] Pearson SJ, Whitaker AF. Footwear in classical ballet: a study of pressure distribution and related foot injury in the adolescent dancer. J Dance Med Sci. 2012;16(2):51-6. PMID 22687718
- [Result] Khan K, Brown J, Way S, Vass N, Crichton K, Alexander R, Baxter A, Butler M, Wark J. Overuse injuries in classical ballet. Sports Med. 1995 May;19(5):341-57. doi: 10.2165/00007256-199519050-00004. PMID 7618011